CLINICAL TRIAL: NCT02100605
Title: A Study to Assess the Speed of Relief From Nasal Congestion With a Hypertonic Saline Nasal Spray (Phytosun Decongestant)
Brief Title: Study on Hypertonic Saline Nasal Spray
Acronym: PhytosunDecon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omega Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014_PhytosunDecon_Cardiff_UK
Record Dates: First submitted 2014-03-21; First posted 2014-04-01 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Nasal Congestion
Keywords: Nasal; Congestion; Decongestion; Hypertonic; Saline solution
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phytosun, decongestant, nasal spray (Active Comparator): Phytosun, decongestant, nasal spray
  Nasal spray 20 ml contains:
  22g/l hypertonic seawater Essential oils of Eucalyptus, Niaouli and Wild menthol
  Instructions for use:
  * Shake the bottle before use
  * Tilt the bottle to one side; press the nozzle firmly for at least one second, repeat until obtaining the 1st spray.
  * Spray in each nostril with the head upright
  Interventions: Device: Phytosun, decongestant, nasal spray
- Isotonic saline, nasal spray (Placebo Comparator): Isotonic saline, nasal spray
  20 ml nasal spray contains Isotonic water solution 0.9% sodium chloride
  Interventions: Device: Phytosun, decongestant, nasal spray

INTERVENTIONS:
Device: Phytosun, decongestant, nasal spray — one time application of the nasal spray

SUMMARY:
Phytosun decongestant nasal spray is a class I medical device registered in the European Union for the treatment of nasal congestion. The spray contains hypertonic seawater and essential oils. The objective of the study is to investigate the effects of a nasal spray, registered as a medical device under the name Phytosun Decongestant in the European Union, on speed of onset of relief of nasal congestion in 50 subjects suffering from nasal congestion associated with common cold.

DETAILED DESCRIPTION:
The study will also include an exploratory assessement of any objective changes in nasal patency by measuring nasal peak inspiratory flow before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged18 years and over
2. Has given written informed consent, and received a copy of their signed consent form prior to any study related procedures
3. Subject considers they are suffering from a common cold of no more than 7 days duration (common cold will be self-diagnosed but all patients will be screened by a doctor and nasal examinations will be performed as needed to establish eligibility of patients for study).
4. Subject on entry to the study has a symptom score of 1 or greater for blocked nose on four point ordinal scale

Exclusion Criteria:

1. Have a known hypersensitivity or are allergic to any component of the test product
2. The subject has a clinically significant cardiovascular, endocrinological, neurological, respiratory, gastrointestinal disease or a history or any current disease that is considered by the investigator as a reason for exclusion e.g. current allergic rhinitis, chronic obstructive pulmonary disease
3. The subject has a severe nasal septal deviation or other condition that could cause nasal obstruction such as the presence of nasal polyps.
4. The subject has had nasal or sinus surgery in the past that in the opinion of the investigator may influence symptom scores
5. The subject has a history of alcohol or other substance abuse in previous year
6. The subject is taking any prescribed medication other than for contraception, that is considered by the investigator as a reason for exclusion e.g. systemic steroids, intranasal medicines, antibiotics.
7. The subject has had common cold or flu like symptoms for more than seven days
8. The subject has recently taken a common cold medicine that in the opinion of the investigator may influence baseline symptom scores (such as nasal decongestants)
9. The subject is a current smoker (more than 2 cigarettes, pipes, cigars a day)
10. The subject is related to any study personnel
11. The subject has received any investigational drug or participated in a clinical trial within 4 weeks of entry to this study
12. The subject is pregnant or lactating -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
assessment of the speed of relief nasal congestion | within 600 seconds after treatment administration
  Subjects will be instructed that the investigator will administer one spray of the treatment into each nasal passage and then start a stop clock. The subject will be asked to stop the clock immediately when they feel any relief of nasal congestion. A sign with the following wording will be placed near the stop-clock.
  STOP THE CLOCK IMMEDIATELY YOU FEEL RELIEF OF NASAL CONGESTION The clock will be stopped after 600 seconds even if the subject does not respond

OTHER OUTCOMES:
nasal peak inspiratory flow | within 20 minutes prior to treatment and within 30 minutes after treatment administration
  The measurement of Peak Nasal Inspiratory Flow (PNIF) (litres/minute) will be performed with the In-Check portable nasal flow meter.
Adverse events monitoring | after all trial related procedures on day 1, which is the day of treatment administration as we only have one visit day.
  Any adverse events (AE) will be documented by asking the subjects to record in the CRF any signs and symptoms after the dose in clinic, Adverse events may also be elicited at the end of the study when the subject is interviewed about their experiences during the study. Adverse events will be recorded in the case report form (CRF) at the final study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Eccles, Professor, Study Director — Common Cold Centre & Healthcare Clinical Trials, Cardiff school of biosciences, Cardiff University; Moutaz SM Jawad, MB ChB FRCP, Principal Investigator — Cardiff University, Cardiff school of biosciences
Locations (1):
- Common Cold Centre & Healthcare Clinical Trials, Cardiff school of biosciences, Cardiff University, Cardiff, United Kingdom